CLINICAL TRIAL: NCT04365192
Title: Comparison of Efficacy of Two Supraglottic Airway Devices: I-gel and the Self-pressurized Air-q in Elderly Patients
Status: Completed | Type: Observational
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Ferda Yilmaz Inal, assistant professor, Istanbul Medeniyet University
Other Study IDs: 2013-KAEK-64
Record Dates: First submitted 2020-04-17; First posted 2020-04-28 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Supraglottic Airway Devices

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- I-gel
  Interventions: Device: I-gel
- Self-pressurized air-Q
  Interventions: Device: Self-pressurized air-Q

INTERVENTIONS:
Device: I-gel — The i-gel airway is a supraglottic airway management device made of thermoplastic elastomer, which is soft, gel-like, and transparent.
  The i-gel has evolved as a device that accurately positions itself over the laryngeal framework, providing a reliable perilaryngeal seal, and therefore no cuff inflation is necessary.
  Groups: I-gel
Device: Self-pressurized air-Q — The self-pressured air-Q is a supraglottic airway management device The intracuff pressure of air-Q dynamically equilibrates with the airway pressure and adjusts to the patient's pharyngeal and periglottic anatomy, potentially providing improved airway fit and seal.
  Groups: Self-pressurized air-Q

SUMMARY:
Supraglottic airway devices with noninflatable cuff have advantages in omitting the cuff pressure monitoring and reducing potential pharyngolaryngeal complications. Typical devices without cuff inflation available are the i-gel™ and the self-pressurized air-Q™ intubating laryngeal airway (air-Q SP).

The i-gel airway is a supraglottic airway management device made of thermoplastic elastomer, which is soft, gel-like, and transparent. It was designed to create a noninflating anatomical seal of the pharyngeal, laryngeal, and perilaryngeal structures while avoiding the compression trauma that can occur with inflatable SADs.

The i-gel has evolved as a device that accurately positions itself over the laryngeal framework, providing a reliable perilaryngeal seal, and therefore no cuff inflation is necessary. Its advantages include easier insertion, minimal risk for tissue compression, and stability after insertion.

The air-Q is a new SAD intended for use as a primary airway and an aid for tracheal intubation in situations of anticipated or unanticipated difficult airways. The intracuff pressure of air-Q dynamically equilibrates with the airway pressure and adjusts to the patient's pharyngeal and periglottic anatomy, potentially providing improved airway fit and seal.

The anatomical and physiological changes that accompany ageing may have a significant influence on the efficacy and safety of SADs. The distinctive features of the air-Q SP and i-gel may lead to a substantial difference in performance in the elderly, and it is planned a head-to-head comparison of these two devices in patients aged between 65 and 85 years.

ELIGIBILITY:
Inclusion Criteria:

* 65-85 years old
* ASA I-III
* Elective urologic surgery
* Mallampati 1-2

Exclusion Criteria:

* BMI>35kg/m2
* Operation time more than 2 hours

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: 65-85 years old patients who undergo urologic surgery
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
Success in first attempt | 3 minutes
  Correct insertion was assessed by proper chest expansion, the presence of a CO2 wave form with a plateau on the capnograph, absence of audible leak, and lack of gastric insufflation.

SECONDARY OUTCOMES:
Fiberoptic view grade | 4 minutes
  Grade 1: whole vocal cords are seen, the epiglottis is not seen at all. Grade 2: larynx plus the posterior surface of epiglottis are seen. Grade 3: the anterior tip of the epiglottis is seen. Grade 4: the anterior tip of the epiglottis is seen and encroaching on the view of vocal cords obstructing <50% of view. Grade 5: the epiglottis is completely obstructing the AQ opening, no view is seen.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medeniyet University, Istanbul, Turkey (Türkiye)